CLINICAL TRIAL: NCT00666887
Title: A Phase III Double-blind, Randomized, Placebo-controlled Trial of Minocycline in Clinically Isolated Syndromes (CIS) and Early Single Relapse Multiple Sclerosis (MS)
Brief Title: Minocycline in Clinically Isolated Syndromes (CIS)
Acronym: MinoCIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Luanne Metz (Other)
Collaborators: Multiple Sclerosis Society of Canada (Other)
Responsible Party: Sponsor-Investigator, Dr. Luanne Metz, Principal Investigator, University of Calgary
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Grant ID # 21569; Health Canada Control #120007 (Other: Health Canada)
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Clinically Isolated Syndromes; Early Single Relapse of Multiple Sclerosis
Keywords: Multiple Sclerosis; Clinically Isolated Syndrome; Minocycline; Placebo
MeSH Terms: conditions — Multiple Sclerosis; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline (Active Comparator): Minocycline 100 mg oral for up to 24 months
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator): Lactose Monohydrate NF (Spray-dried) 235 mg/cap Magnesium Stearate NF 1 mg/cap Croscarmellose Sodium NF 4 mg/cap Stearic Acid 10 mg/cap Placebo CAP Lt orange OP-Purple OP (APO 100)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minocycline — 100 mg twice daily to be taken for up to 2 years
  Other Names: MINOCIN; Minocycline Hydrochloride
  Arms: Minocycline
Drug: Placebo — placebo twice daily for 2 years
  Arms: Placebo

SUMMARY:
The aim of the trial is to demonstrate that 100 mg of oral minocycline twice daily reduces the conversion of CIS to McDonald Criteria MS (McDMS) by an absolute 25% as compared to placebo, over a 6 month follow-up period (primary outcome).

A key secondary outcome is to confirm that this early treatment benefit is maintained at two years.

DETAILED DESCRIPTION:
* Minocycline 100 mg bid orally compared to identical placebo
* Clinically Isolated Syndrome (CIS): Patients with a first clinical demyelinating event suggestive of multiple sclerosis (At baseline participants may meet 2010 McDonald diagnostic criteria for MS, but not 2005 criteria)
* Men and women, aged 18-60y, first event within the previous 180 days; brain magnetic resonance imaging (MRI) with at least two brain T2 lesions which are at least 3 mm in diameter, and at least one of which is ovoid or periventricular or infratentorial.
* Up to 24 months of study drug (Up to 12 months of study drug for patients recruited after December 31, 2012)
* Patients will be discontinued from the study when they convert to McDMS based on the 2005 McDonald definition.
* 12 Canadian MS Clinics
* A total of 154 patients will be randomized. Because 30% of screened patients with CIS who are clinically eligible are not expected to meet the MRI criteria for inclusion, up to 280 patients will be screened.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years.
* First focal clinical episode suggestive of demyelinating disease within the previous 180 days (measured from onset of the first symptom to treatment start), based on the appearance of a neurological abnormality, present for at least 24 hours.
* Objective clinical evidence must be present or documented. Patients will be included irrespective of whether the first clinical demyelinating episode was monosymptomatic (i.e. clinical evidence of a single lesion) or polysymptomatic (i.e. clinical evidence of more than one lesion).
* At least two lesions on the T2-weighted brain MRI* scan at least one of which is ovoid or periventricular or infratentorial. MRI eligibility will be determined centrally by the UBC MS/MRI Research Group.*One lesion on spinal MRI may substitute for one brain lesion as per the 2005 McDonald Criteria.
* Sexually active women of child-bearing potential must agree to use adequate contraception.
* Written informed consent

Exclusion Criteria:

* Any disease other than MS that could better explain the patient's signs and symptoms.
* Any previous clinical event reasonably attributable to acute demyelination, regardless of whether medical attention was obtained.
* Complete transverse myelitis or bilateral optic neuritis. A waiver can be obtained for bilateral optic neuritis but must be obtained prior to randomization. Waivers must be approved by 3 neurologists including a member of the Clinical Eligibility / Endpoint Committee, a member of the DSMC, and by an experienced MS neurophthalmologist.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2009-01; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To demonstrate that 100 mg of oral minocycline twice daily reduces the conversion of CIS to McDonald Criteria MS (McDMS) by an absolute 25% as compared to placebo, over a 6 month follow-up period. | 6 Months

SECONDARY OUTCOMES:
To confirm that this early treatment benefit is maintained at two years. | 2 years
Change in T2 lesion volume | 6 months and 24 months
Cumulative number of enhancing T1 lesions | 6 months and 24 months
cumulative combined unique lesions (new enhancing T1-weighted lesions plus new and enlarging T2 lesions, without lesion double counting) | 6 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Luanne Metz, MD, Principal Investigator — University of Calgary
Locations (12):
- Canada (12):
  - University of Calgary, Calgary Health Region, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Fraser Health Multiple Sclerosis Clinic, Burnaby, British Columbia
  - UBC Hospital, Vancouver, British Columbia
  - MS Research Unit, Health Sciences Centre, Winnipeg, Manitoba
  - Dalhousie MS Research Unit, Halifax, Nova Scotia
  - MS Clinic, London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Multiple Sclerosis Research Clinic, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Clinique Neuro Rive-Sud, Greenfield Park, Quebec
  - CHUM Notre-Dame, Montreal, Quebec
  - CHAUQ Enfant-Jesus, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No
Consent to share IPD was not obtained from subjects so data cannot be shared except amongst investigators.

REFERENCES:
- [Derived] Camara-Lemarroy C, Metz L, Kuhle J, Leppert D, Willemse E, Li DK, Traboulsee A, Greenfield J, Cerchiaro G, Silva C, Yong VW. Minocycline treatment in clinically isolated syndrome and serum NfL, GFAP, and metalloproteinase levels. Mult Scler. 2022 Nov;28(13):2081-2089. doi: 10.1177/13524585221109761. Epub 2022 Jul 18. PMID 35848622
- [Derived] Metz LM, Li DKB, Traboulsee AL, Duquette P, Eliasziw M, Cerchiaro G, Greenfield J, Riddehough A, Yeung M, Kremenchutzky M, Vorobeychik G, Freedman MS, Bhan V, Blevins G, Marriott JJ, Grand'Maison F, Lee L, Thibault M, Hill MD, Yong VW; Minocycline in MS Study Team. Trial of Minocycline in a Clinically Isolated Syndrome of Multiple Sclerosis. N Engl J Med. 2017 Jun 1;376(22):2122-2133. doi: 10.1056/NEJMoa1608889. PMID 28564557
- [Derived] Kang H, Metz LM, Traboulsee AL, Eliasziw M, Zhao GJ, Cheng Y, Zhao Y, Li DK; Minocycline in CIS Study Group. Application and a proposed modification of the 2010 McDonald criteria for the diagnosis of multiple sclerosis in a Canadian cohort of patients with clinically isolated syndromes. Mult Scler. 2014 Apr;20(4):458-63. doi: 10.1177/1352458513501230. Epub 2013 Aug 22. PMID 23970502